CLINICAL TRIAL: NCT06906406
Title: Health-Related Quality of Life in Children and Adolescents With Clubfoot. A Prospective Observational Study
Brief Title: Health-Related Quality of Life in Children and Adolescents With Clubfoot
Status: Recruiting | Type: Observational
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 1000323
Record Dates: First submitted 2025-03-07; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Clubfoot; Children; HRQOL (Health Related Quality Of Life)
Keywords: HRQoL; PedsQL; Children; Clubfoot; Ponseti
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This prospective cohort study aims to evaluate the health-related quality of life (HRQoL) in children aged 2 to 15 years with congenital clubfoot, treated primarily according to the Ponseti method. The study will assess HRQoL using the Pediatric Quality of Life Inventory (PedsQL 4.0) and clinical outcomes using the PBS Clubfoot Score (PBS). Participants will be followed for 2 and 5 years to evaluate changes in HRQoL and clinical function. The primary objective is to understand the long-term impact of clubfoot and its treatment on patients' physical, emotional, and social well-being.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 to 15 years diagnosed with congenital clubfoot.
* Undergoing treatment or follow-up at Drammen Hospital.
* Both unilateral and bilateral cases included.
* Written informed consent from parents or legal guardians.

Exclusion Criteria:

* Concurrent severe medical or psychological conditions affecting outcomes.
* Lack of written informed consent.
* Incomplete or missing data for PedsQL or PBS assessments.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study investigates the impact of congenital clubfoot and its treatment on the health-related quality of life (HRQoL) in children using a prospective cohort design. The participants will be evaluated using the Pediatric Quality of Life Inventory (PedsQL 4.0) to assess HRQoL and the PBS Clubfoot Score (PBS) for clinical outcomes. Assessments will occur at baseline, 2 years, and 5 years post-treatment initiation. Data collection will include clinical evaluations, standardized HRQoL questionnaires, and Visual Analogue Scale (VAS) assessments for pain and satisfaction. The findings will help optimize treatment protocols for clubfoot by providing comprehensive insights into how different treatment methods impact children's quality of life.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
HRQoL Score | Baseline, then at every follow-up over the study period of a total of 5 years.
  Health-Related Quality-of-Life (HRQoL) score as measured by The Pediatric Quality of Life Inventory™ (PedsQL) 4.0, assessing physical, emotional, social, and school functioning. Scored on a scale from 0 to 100, with higher scores indicating better HRQoL.

SECONDARY OUTCOMES:
PBS Clubfoot Score | Baseline, then at every follow-up over the study period of a total of 5 years.
  The PBS (Ponseti, Barlow, and Stagnara) Clubfoot Score assesses clinical function, including foot shape, range of motion, and muscle balance. The score ranges from 7 to 18 points, in which a low score indicates good function, and a high score indicates poor function.
Pain Assessment | Baseline, then at every follow-up over the study period of a total of 5 years.
  Pain Assessment: Visual Analogue Scale (VAS) score ranging from 0 (no pain) to 100 (worst pain imaginable).
Satisfaction Assessment | Baseline, then at every follow-up over the study period of a total of 5 years.
  Satisfaction Assessment: Visual Analogue Scale (VAS) score for patient and parent satisfaction with treatment outcomes, ranging from 0 (not satisfied) to 100 (completely satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Vestreviken, Drammen, Buskerud, Norway

IPD SHARING:
Plan to Share IPD: No